CLINICAL TRIAL: NCT06527911
Title: A Randomized Controlled Trial of the Sagittal Alignment Difference Between Mako Robotic Total Knee Arthroplasty and Manual Total Knee Arthroplasty
Brief Title: A Randomized Controlled Trial of the Sagittal Alignment Difference Between Mako Robotic TKA and Manual TKA
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Jiafeng Yi, Resident doctor, Chinese PLA General Hospital
Other Study IDs: 2023KY023-KS001
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Arthroplasty; Replacement; Knee; Osteoarthritis; Robotic Surgical Procedures
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mako robot assisted TKA: Patients with osteoarthritis (OA) who underwent Mako robot-assisted TKA at the Chinese PLA General Hospital between September 2024 and September 2026.
- Manual TKA: Patients with OA who underwent manual TKA at the Chinese PLA General Hospital between September 2024 and September 2026.

SUMMARY:
As China transitions into an aging society, the proportion of the elderly population is escalating, with a corresponding rise in the number of patients with knee joint diseases. Total knee arthroplasty stands as an effective treatment for joint disorders, effectively reducing knee pain, restoring functionality, and enhancing quality of life. The objectives of total knee arthroplasty are to relieve pain, restore function, and ensure a long-lasting implant. In recent years, technological advancements have integrated robotic assistance into total knee arthroplasty (TKA), aiding surgeons in planning and executing more accurate surgical plans, significantly enhancing precision and post-operative outcomes. However, the Mako mechanical axis alignment demonstrated during the Mako robot-assisted TKA procedure does not correspond to the actual straightening of the lower limb, and discrepancies may exist in sagittal alignment between Mako-assisted and manual TKA procedures, necessitating adjustments by surgeons based on their experience. Consequently, there is an urgent need to develop a mathematical formula that quantifies these differences to guide intraoperative alignment. Additionally, the Mako-assisted TKA femoral prosthesis exhibits a head-lowering issue, and differences exist in the posterior slope angle of the tibial plateau compared to manual TKA, necessitating further comparative analysis to draw definitive conclusions. This study will be carried out at the People's Liberation Army General Hospital, with an anticipated enrollment of approximately 100 participants.

DETAILED DESCRIPTION:
I. Clinical Research Background As China transitions into an aging society, the proportion of the elderly population is escalating, with a corresponding rise in the number of patients with knee joint diseases. Total knee arthroplasty stands as an effective treatment for joint disorders, effectively reducing knee pain, restoring functionality, and enhancing quality of life. The objectives of total knee arthroplasty are to relieve pain, restore function, and ensure a long-lasting implant. In recent years, technological advancements have integrated robotic assistance into total knee arthroplasty (TKA), aiding surgeons in planning and executing more accurate surgical plans, significantly enhancing precision and post-operative outcomes. However, the Mako mechanical axis alignment demonstrated during the Mako robot-assisted TKA procedure does not correspond to the actual straightening of the lower limb, and discrepancies may exist in sagittal alignment between Mako-assisted and manual TKA procedures, necessitating adjustments by surgeons based on their experience. Consequently, there is an urgent need to develop a mathematical formula that quantifies these differences to guide intraoperative alignment. Additionally, the Mako-assisted TKA femoral prosthesis exhibits a head-lowering issue, and differences exist in the posterior slope angle of the tibial plateau compared to manual TKA, necessitating further comparative analysis to draw definitive conclusions.

II. Content of Clinical Trials (I) Overall Design and Sample Size This study is a prospective clinical investigation, encompassing two groups: ① the Mako robot-assisted TKA group: patients with osteoarthritis (OA) who underwent Mako robot-assisted TKA at the Chinese PLA General Hospital between September 2024 and September 2026; and ② the manual TKA group: patients with OA who underwent manual TKA at the same hospital between September 2024 and September 2026.

(II) Randomization and Control in the Trial Randomized Controlled Trial (III) Content This clinical study aims to compare the differences between the extension demonstrated during Mako robot-assisted TKA surgery and the actual postoperative extension, proposing a mathematical formula to reflect these discrepancies. Through the validation of intraoperative and postoperative data, the study aims to guide the extension during Mako-assisted TKA. Additionally, In Mako-assisted TKA, there is a femoral prosthesis bowing down issue, and the posterior inclination angle of the tibial plateau differs from that of manual TKA. Consequently, the sagittal femoral bowing down angle and posterior inclination angle of the tibial plateau were compared between robot-assisted TKA and manual TKA to verify the differences between the groups.This study was conducted at the Joint Surgery Department of the Chinese PLA General Hospital, with participants meeting inclusion criteria and not violating exclusion criteria, and having signed informed consent forms approved by the ethics committee.

III: Trial Procedure (I) Participant Enrollment Physicians selected osteoarthritis (OA) patients who underwent total knee arthroplasty (TKA) at our hospital from September 2024 to September 2026, and screened them based on inclusion and exclusion criteria. If a patient met the inclusion criteria, the details of the research project were thoroughly explained to them, and they were required to sign the relevant informed consent form.

(II) Methodology A clinical study was conducted at the Joint Surgery Department of the Chinese PLA General Hospital from September 2024 to September 2026, involving 50 patients each undergoing Mako robot-assisted TKA and manual TKA (Stryker Triathlon prosthesis). Basic patient information, including ID number, name, gender, age, height, and weight, was recorded. Preoperative and postoperative full-length lateral radiographs of the lower limbs, bilateral knee joint lateral radiographs, and sagittal EOS of the lower limbs were taken for all patients. An experienced researcher measured the posterior slope angle of the tibial plateau preoperatively and postoperatively using the Mako robot-assisted TKA, as well as the extension angle displayed by the Mako at the end of the TKA procedure. Based on the differences preoperatively and postoperatively in the 50 cases of Mako robot-assisted TKA, a mathematical formula reflecting extension was proposed and validated. Preoperative and postoperative coronal HKA, LDFA, and MPTA measurements were taken for both Mako robot-assisted TKA and manual TKA; preoperative and postoperative sagittal measurements of the posterior slope angle of the tibial plateau; and postoperative femoral prosthesis head tilt angle were recorded, and statistical analysis was conducted to compare the sagittal angle differences between Mako robot-assisted and manual TKA.

(III) Clinical Evaluation Indices (1) Primary Outcome Measures:

1. The extension angle displayed by the Mako robot at the conclusion of the Mako-assisted Total Knee Arthroplasty (TKA) procedure;
2. Sagittal plane femoral anterior arch angle;
3. Preoperative and postoperative coronal hip-knee-ankle (HKA) angles, lateral distal femoral angle (LDFA), and medial proximal tibial angle (MPTA) in Mako robot-assisted TKA and manual TKA;
4. Preoperative and postoperative sagittal measurement of the tibial plateau posterior slope angle; postoperative femoral prosthesis head-down angle.

(2) Secondary Observational Indicators

1. Basic demographic data of the patients.

* Statistical Analysis Methods All results were computed using SPSS 26.0. A comprehensive enumeration of the collected data will be presented, followed by a descriptive summary of the data. Categorical variables will be summarized using frequencies and percentages, while continuous variables will be summarized by the number of subjects at each evaluation time point, mean values, mean differences relative to baseline values (where appropriate), medians, standard deviations, 95% confidence intervals, minimum values, and maximum values.

Prior to database lock, the definitive statistical analysis plan will be established, and the pertinent clinical and statistical personnel will document their decisions regarding the inclusion or exclusion of data from each subject.

ELIGIBILITY:
Inclusion Criteria:

1. The age ranged from 18 to 80 years old;
2. OA patients who underwent Mako robot assisted TKA and manual TKA (Stryker Triathlon prosthesis) in the Department of joint surgery of the PLA General Hospital from September 2024 to September 2026;
3. All patients were required to take full-length anteroposterior and lateral radiographs of lower limbs, anteroposterior and lateral radiographs of both knees, and lower limb sagittal EOS before and after surgery;
4. Physical and mental health, able to participate in and cooperate with the test;
5. Patients are willing to participate in the study and sign written informed consent.

Exclusion Criteria:

1. People unable to conduct EOS inspection;
2. Combined with knee meniscus injury, anterior cruciate ligament injury and other diseases that may affect the sagittal force line of the knee joint
3. Combined with other diseases that may affect the study
4. Patients refused to use their imaging data and knee score for this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: OA patients who underwent Mako robot assisted TKA and manual TKA (Stryker Triathlon prosthesis) in the Department of joint surgery of the PLA General Hospital from September 2024 to September 2026 were screened.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
The extension angle displayed by the Mako robot at the conclusion of the Mako-assisted Total Knee Arthroplasty (TKA) procedure | From admission to discharge, up to 1 week
Sagittal plane femoral anterior arch angle | From admission to discharge, up to 1 week
Preoperative and postoperative coronal hip-knee-ankle (HKA) angles, lateral distal femoral angle (LDFA), and medial proximal tibial angle (MPTA) in Mako robot-assisted TKA and manual TKA | From admission to discharge, up to 1 week
Preoperative and postoperative sagittal measurement of the tibial plateau posterior slope angle; postoperative femoral prosthesis head-down angle | From admission to discharge, up to 1 week

SECONDARY OUTCOMES:
Basic demographic profile of the patient | From admission to discharge, up to 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chai, doctorate, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China